CLINICAL TRIAL: NCT00789035
Title: A Phase IIb, Randomized, Parallel Group Safety, Efficacy, and Pharmacokinetics Study of BI 10773 (5 mg, 10 mg and 25 mg) Administered Orally Once Daily Over 12 Weeks Compared Double Blind to Placebo, as Monotherapy, With an Additional Open-label Metformin Arm in Type 2 Diabetic Patients With Insufficient Glycemic Control
Brief Title: 12 Weeks Treatment With 3 Different Doses of BI 10773 in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1245.9; EudraCT No 2008-000640-14
Record Dates: First submitted 2008-10-13; First posted 2008-11-11 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Metformin

INTERVENTIONS:
Drug: BI 10773
Drug: placebo
Drug: metformin

SUMMARY:
The objective is to investigate the efficacy, safety and pharmacokinetics of three different doses of BI 10773 compared to placebo given for 12 weeks in patients with type 2 diabetes mellitus with insufficient glycemic control. In addition an open-label metformin arm will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a diagnosis of type 2 diabetes mellitus
* either treatment-naïve or on a maximum of 1 oral antidiabetic therapy on a stable dose for the10 weeks prior to screening
* HbA1c ≥6.5 to ≤9.0% and for treatment-naïve patients:HbA1c >7.0 to ≤10.0%
* HbA1c >7.0 to ≤10.0% at Visit 2 (start of run-in) for all patients
* Age between 18 and 80 years
* BMI less than 40 kg/m2
* Signed and dated informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion Criteria:

1. Myocardial infarction, stroke or TIA within 6 months prior to informed consent
2. Impaired hepatic function
3. Renal insufficiency or impaired renal function
4. Disease of central nervous system, or psychiatric disorders or clinically relevant neurologic disorders that may interfere with trial participation
5. Chronic or clinically relevant acute infections
6. Current or chronic urogenital tract infection determined by medical history
7. History of clinically relevant allergy/hypersensitivity
8. Treatment with glitazones, GLP-1 analogues or insulin within 3 months prior to informed consent
9. Treatment with anti obesity drugs
10. Current treatment with systemic steroids
11. Alcohol abuse
12. Treatment with an investigational drug within 2 months prior to informed consent
13. known intolerance to metformin
14. Dehydration
15. Unstable or acute CHF
16. Acute or chronic acidosis
17. Hereditary galactose intolerance
18. Woman of child bearing potential who are nursing or pregnant or not practicing an acceptable method of birth control

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (74):
- Argentina (10):
  - 1245.9.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54007 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54008 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54009 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54010 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.9.54004 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1245.9.54003 Boehringer Ingelheim Investigational Site, Mendoza
  - 1245.9.54005 Boehringer Ingelheim Investigational Site, Salta
  - 1245.9.54006 Boehringer Ingelheim Investigational Site, Salta
- Croatia (5):
  - 1245.9.38504 Boehringer Ingelheim Investigational Site, Karlovac
  - 1245.9.38503 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1245.9.38506 Boehringer Ingelheim Investigational Site, Osijek
  - 1245.9.38505 Boehringer Ingelheim Investigational Site, Varaždin
  - 1245.9.38501 Boehringer Ingelheim Investigational Site, Zagreb
- Estonia (3):
  - 1245.9.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.9.37202 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.9.37203 Boehringer Ingelheim Investigational Site, Tallinn
- Germany (8):
  - 1245.9.49007 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1245.9.49001 Boehringer Ingelheim Investigational Site, Erlangen
  - 1245.9.49004 Boehringer Ingelheim Investigational Site, Hamburg
  - 1245.9.49005 Boehringer Ingelheim Investigational Site, Hamburg
  - 1245.9.49002 Boehringer Ingelheim Investigational Site, Melsungen
  - 1245.9.49008 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1245.9.49003 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1245.9.49006 Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
- Italy (5):
  - 1245.9.39006 Boehringer Ingelheim Investigational Site, Genova
  - 1245.9.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1245.9.39003 Boehringer Ingelheim Investigational Site, Pisa
  - 1245.9.39004 Boehringer Ingelheim Investigational Site, Siena
  - 1245.9.39005 Boehringer Ingelheim Investigational Site, Treviso
- Lithuania (2):
  - 1245.9.37002 Boehringer Ingelheim Investigational Site, Klaipėda
  - 1245.9.37001 Boehringer Ingelheim Investigational Site, Vilnius
- Romania (4):
  - 1245.9.40003 Boehringer Ingelheim Investigational Site, Brasov
  - 1245.9.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.9.40004 Boehringer Ingelheim Investigational Site, Galati
  - 1245.9.40005 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Russia (7):
  - 1245.9.70002 Boehringer Ingelheim Investigational Site, Kazan'
  - 1245.9.70003 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 1245.9.70004 Boehringer Ingelheim Investigational Site, Petrozavodsk
  - 1245.9.70005 Boehringer Ingelheim Investigational Site, Smolensk
  - 1245.9.70006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1245.9.70007 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1245.9.70001 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Slovakia (4):
  - 1245.9.62002 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.9.62003 Boehringer Ingelheim Investigational Site, Lučenec
  - 1245.9.62004 Boehringer Ingelheim Investigational Site, Nové Mesto nad Váhom
  - 1245.9.62001 Boehringer Ingelheim Investigational Site, Prievidza
- South Korea (9):
  - 1245.9.82006 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.9.82008 Boehringer Ingelheim Investigational Site, Goyang
  - 1245.9.82007 Boehringer Ingelheim Investigational Site, Incheon
  - 1245.9.82002 Boehringer Ingelheim Investigational Site, Pucheon
  - 1245.9.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.9.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.9.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1245.9.82009 Boehringer Ingelheim Investigational Site, Suwon
  - 1245.9.82003 Boehringer Ingelheim Investigational Site, Uijeongbu-si
- Sweden (5):
  - 1245.9.46003 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1245.9.46004 Boehringer Ingelheim Investigational Site, Härnösand
  - 1245.9.46005 Boehringer Ingelheim Investigational Site, Lund
  - 1245.9.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1245.9.46002 Boehringer Ingelheim Investigational Site, Västerås
- Taiwan (7):
  - 1245.9.88605 Boehringer Ingelheim Investigational Site, Changhua
  - 1245.9.88607 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1245.9.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 1245.9.88606 Boehringer Ingelheim Investigational Site, Tainan
  - 1245.9.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.9.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 1245.9.88602 Boehringer Ingelheim Investigational Site, Taoyuan District
- Ukraine (5):
  - 1245.9.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.9.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.9.38002 Boehringer Ingelheim Investigational Site, Odesa
  - 1245.9.38001 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 1245.9.38005 Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Riggs MM, Staab A, Seman L, MacGregor TR, Bergsma TT, Gastonguay MR, Macha S. Population pharmacokinetics of empagliflozin, a sodium glucose cotransporter 2 inhibitor, in patients with type 2 diabetes. J Clin Pharmacol. 2013 Oct;53(10):1028-38. doi: 10.1002/jcph.147. Epub 2013 Aug 13. PMID 23940010

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive Placebo in tablets matching the Empagliflozin tablets in appearance once daily.
- Empagliflozin 5 mg: Patients receive 5 mg Empagliflozin in tablets once daily.
- Empagliflozin 10 mg: Patients receive 10 mg Empagliflozin in tablets once daily.
- Empagliflozin 25 mg: Patients receive 25 mg Empagliflozin in tablets once daily.
- Metformin OL: Patients were to take a open-label (OL) dose of 500 mg Metformin twice daily for the first 4 weeks. For the remaining 8 weeks, if the fasted blood glucose values were above 110 mg/dL (6.1 mmol/L), the dose was to be increased to 2 x 500 mg tablets twice daily or up to the maximum tolerated.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Started | 82 | 81 | 81 | 82 | 80
Completed | 76 | 74 | 80 | 81 | 74
Not Completed | 6 | 7 | 1 | 1 | 6
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 3
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Not completed — Other reason not defined above | 2 | 3 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisting of all randomised patients who were treated with at least 1 dose of study drug.
Groups:
- Metformin OL: Patients were to take a dose of 500 mg Metformin (open-label) twice daily for the first 4 weeks. For the remaining 8 weeks, if the fasted blood glucose values were above 110 mg/dL (6.1 mmol/L), the dose was to be increased to 2 x 500 mg tablets twice daily or up to the maximum tolerated.
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL | Total
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.2) | 58.4 (9.7) | 58.2 (9.9) | 56.4 (10.3) | 57.0 (8.9) | 57.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 41 | 41 | 41 | 195
  Male | 45 | 46 | 40 | 41 | 39 | 211

OUTCOME MEASURES:

1. Primary Outcome: Change of Glycosilated Haemoglobin A1c (HbA1c) From Baseline After 12 Weeks of Treatment
Description: Change of HbA1c from baseline after 12 weeks of treatment.
  Note, adjusted means are presented. For the placebo and empa groups, measured values presented are for the model including only these treatment groups, for the metformin group the measured values presented are for the model including only placebo and metformin groups.
Time Frame: Baseline and 12 weeks
Population: The full analysis set (FAS) consists of all randomised patients who were treated with at least 1 dose of study drug and had a baseline measurement of the primary endpoint. Modified last observation carried forward was used as the imputation method (LOCF).
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80
percentage of HbA1c | 0.09 (0.09) | -0.43 (0.09) | -0.48 (0.09) | -0.63 (0.09) | -0.75 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — No formal testing so adjustment for multiple comparisons was not necessary; Based on ANCOVA with terms for baseline, treatment, number of previous anti-diabetic medications and country; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.74 to -0.29], Standard Error of Mean 0.11 — Difference calculated as empa 5mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — No formal testing so adjustment for multiple comparisons was not necessary; Based on ANCOVA with terms for baseline, treatment, number of previous anti-diabetic medications and country; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.80 to -0.35], Standard Error of Mean 0.11 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — No formal testing so adjustment for multiple comparisons was not necessary; Based on ANCOVA with terms for baseline, treatment, number of previous anti-diabetic medications and country; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.94 to -0.50], Standard Error of Mean 0.11 — Difference calculated as empa 25mg minus placebo

2. Secondary Outcome: Change of FPG From Baseline After 12 Weeks of Treatment
Description: Change of Fasting Plasma Glucose (FPG) from baseline after 12 weeks of treatment. Results presented stem from a repeated measures analysis.
  Note, adjusted means are presented. For the placebo and empa groups, measured values presented are for the model including only these treatment groups, for the metformin group the measured values presented are for the model including only placebo and metformin groups.
Time Frame: Baseline and 12 weeks
Population: FAS (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 80 | 80 | 82 | 80
mg/dL | 0.79 (3.54) | -23.26 (3.59) | -28.92 (3.59) | -31.08 (3.59) | -29.96 (4.02)

3. Secondary Outcome: Change of HbA1c From Baseline Over Time
Description: Change of HbA1c from baseline over time. Results presented stem from a repeated measures analysis.
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS, classical last observation carried forward (CLOCF) was used as the imputation method.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80
percentage of HbA1c
  Week 4 | -0.01 (0.06) | -0.27 (0.06) | -0.24 (0.06) | -0.39 (0.06) | -0.26 (0.07)
  Week 8 | 0.04 (0.07) | -0.43 (0.08) | -0.53 (0.08) | -0.58 (0.07) | -0.59 (0.08)
  Week 12 | 0.07 (0.08) | -0.47 (0.08) | -0.53 (0.08) | -0.66 (0.08) | -0.78 (0.08)

4. Secondary Outcome: Proportion of Patients Who Achieve an HbA1c ≤7.0% After 12 Weeks of Treatment
Description: Results for HbA1c categories at week 12 (Proportion of patients with HbA1c less than equal to 7%).
Time Frame: 12 weeks
Population: FAS (CLOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80
percentage of participants | 22.0 | 33.3 | 29.6 | 45.1 | 45.0

5. Secondary Outcome: Proportion of Patients Who Achieve an HbA1c Lowering of at Least 0.5% After 12 Weeks of Treatment
Description: Results for HbA1c categories at week 12 (Proportion of patients with HbA1c lowered at least 0.5%).
Time Frame: 12 weeks
Population: FAS (CLOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80
percentage of participants | 25.6 | 46.9 | 59.3 | 59.8 | 71.3

6. Secondary Outcome: Change From Baseline to Week 12 in Fasting Plasma Insulin (FPI)
Description: Results for change of FPI from baseline at week 12 based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU/L
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 70 | 69 | 70 | 77 | 68
mU/L | -0.95 (0.53) | -0.90 (0.53) | -1.02 (0.53) | -0.90 (0.50) | -0.01 (0.54)

7. Secondary Outcome: Change in Homeostasis Model Assessment Index for Insulin Resistance (HOMA-IR)
Description: HOMA-IR (to assess insulin resistance) is defined as (FPI x FPG)/22.5. Results based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU/L x mmol/L
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 70 | 69 | 70 | 77 | 68
mU/L x mmol/L | -0.19 (0.26) | -0.85 (0.27) | -0.83 (0.26) | -0.79 (0.25) | -0.37 (0.27)

8. Secondary Outcome: Change in Homeostasis Model Assessment Index for Beta Cell Function (HOMA-%B)
Description: HOMA-%B (to assess insulin beta cell function) is defined as (20 x FPI)/(FPG-3.5). Results are based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU / mmol
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 70 | 69 | 70 | 77 | 68
mU / mmol | -5.20 (2.56) | 4.22 (2.57) | 1.09 (2.54) | 2.13 (2.43) | 6.69 (2.58)

9. Secondary Outcome: Change of Body Weight After 12 Weeks of Treatment
Description: Results for change of body weight after 12 weeks of treatment based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Metformin OL
Number analyzed (Participants) | 82 | 81 | 81 | 82 | 80
kg | -0.75 (0.26) | -1.81 (0.26) | -2.33 (0.26) | -2.03 (0.26) | -1.32 (0.26)

10. Secondary Outcome: Trough Concentrations of Empagliflozin in Plasma
Description: Pre-dose (within 30 minutes before dosing) trough concentrations of Empagliflozin in plasma
Time Frame: Days 28, 56 and 84
Population: All patients who received at least one dose of Empagliflozin and have some Pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 70 | 77 | 77
nmol/L
  Day 28 (N=67, 75, 77) | 31.6 (158) | 61.7 (169) | 117 (154)
  Day 56 (N=69, 73, 75) | 20.3 (128) | 51.6 (190) | 127 (140)
  Day 84 (N=70, 77, 75) | 22.9 (132) | 55.3 (156) | 118 (179)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last intake of study medication, up to 121 days
Groups:
- Empagliflozin 10 mg qd: Patients receive 10 mg Empagliflozin in tablets once daily.
- Empagliflozin 25 mg qd: Patients receive 25 mg Empagliflozin in tablets once daily.
Arm/Group | Placebo | Empagliflozin 5 mg | Empagliflozin 10 mg qd | Empagliflozin 25 mg qd | Metformin OL
Serious Adverse Events (participants affected / at risk) | 0/82 | 2/81 | 0/81 | 1/82 | 3/80
Other Adverse Events (participants affected / at risk) | 1/82 | 3/81 | 5/81 | 1/82 | 7/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Empagliflozin 5 mg (N=81) | Empagliflozin 10 mg qd (N=81) | Empagliflozin 25 mg qd (N=82) | Metformin OL (N=80)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Empagliflozin 5 mg (N=81) | Empagliflozin 10 mg qd (N=81) | Empagliflozin 25 mg qd (N=82) | Metformin OL (N=80)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 7
Thirst (General disorders) | 0 | 2 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.